CLINICAL TRIAL: NCT04933266
Title: Ultrasound-guided Subpectoral Plexus Block With Multi-level Thoracic Paravertebral Block for Surgical Anaesthesia During Primary Breast Cancer Surgery: A Prospective Randomized Double-blind Trial
Brief Title: Subpectoral Plexus Block With Multi-level TPVB for Surgical Anesthesia During Primary Breast Cancer Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Manoj K Karmakar, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021.248-T mTPVB SPPB Ver 2
Record Dates: First submitted 2021-06-17; First posted 2021-06-21 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Subpectoral plexus block; Thoracic paravertebral block; Primary breast cancer surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Pharmaceutical Preparations; Levobupivacaine

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to received either 10ml of 0.25% levobupivacaine (Group LD) or 20ml of 0.25% levobupivacaine (Group HD). The randomization sequence will be generated using an online randomization software (www.randomization.com). The randomization sequence will be assigned as 1=low dose 10ml (Group LD) and 2=high dose 20ml (Group HD). The group allocation will be prepared by a computer officer (third party) in the Department of Anaesthesia & Intensive Care of the Chinese University of Hong Kong.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients in both study groups will not be able to know the dosage they will receive during the block and therefore will be blinded to group allocation. The "outcome assessor" (research nurse) will not be presented in the procedure room during block placement and thus will also be blinded to group allocation. The anesthesiologist (principal investigator) performing the allocated block will take no further part in the study after block placement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose (Active Comparator): After three injections of thoracic paravertebral block at T2, T4, T6 (a total of 21ml of 0.5% levobupivacaine with 1:200,000 adrenaline) under ultrasound guidance, patients will be put in supine position with ipsilateral arm and elbow flexed. Ultrasound scan will be performed below collarbone region, 5ml of 0.25% levobupivacaine will be injected in the first plane between pectoralis major and minor. Then under direct ultrasound visualization, the remaining 5ml of 0.25% levobupivacaine will be injected between the second plane of pectoralis minor and serratus anterior muscle (a total of 10ml will be given).
  Interventions: Procedure: Subpectoral plexus block (low dose)
- High dose (Active Comparator): After three injections of thoracic paravertebral block at T2, T4, T6 (a total of 21ml of 0.5% levobupivacaine with 1:200,000 adrenaline) under ultrasound guidance, patients will be put in supine position with ipsilateral arm and elbow flexed. Ultrasound scan will be performed below collarbone region, 10ml of 0.25% levobupivacaine will be injected in the first plane between pectoralis major and minor. Then under direct ultrasound visualization, the remaining 10ml of 0.25% levobupivacaine will be injected between the second plane of pectoralis minor and serratus anterior muscle (a total of 20ml will be given).
  Interventions: Procedure: Subpectoral plexus block (High dose)

INTERVENTIONS:
Procedure: Subpectoral plexus block (low dose) — It is one type of peripheral nerve blocks for surgery over the chest. Patients will have an ultrasound scan and nerve block with local anesthetic (LA) agent (0.25% levobupivacaine 10ml) injected 2 target sites through one skin puncture. One at the myofascial plane between the pectoralis major and minor (5ml of LA) and then under direct ultrasound visualization, the needle will be redirected and the remaining 5ml of LA will be injected at the plane between the pectoralis minor and the serratus anterior muscle, close to the origin of thoracoacromial artery from the axillary artery at the level of the third rib.
  Other Names: Drug (0.25% Chirocaine)
  Arms: Low dose
Procedure: Subpectoral plexus block (High dose) — It is one type of peripheral nerve blocks for surgery over the chest. Patients will have an ultrasound scan and nerve block with local anesthetic (LA) agent (0.25% levobupivacaine 20ml) injected 2 target sites through one skin puncture. One at the myofascial plane between the pectoralis major and minor (10ml of LA) and then under direct ultrasound visualization, the needle will be redirected and the remaining 10ml of LA will be injected at the plane between the pectoralis minor and the serratus anterior muscle, close to the origin of thoracoacromial artery from the axillary artery at the level of the third rib.
  Other Names: Drug (0.25% Chirocaine)
  Arms: High dose

SUMMARY:
The objective of this study is to compare two different doses of local anesthetics (10ml vs 20ml of 0.25% levobupivacaine) for subpectoral plexus block (SPPB) in addition to ultrasound guided multi-level of thoracic paravertebral block (m-TPVB) for surgical anaesthesia for major primary breast cancer surgery.

DETAILED DESCRIPTION:
Primary breast cancer surgery is one of the most commonly performed surgeries worldwide. It is associated with significant acute postoperative pain and a high incidence of chronic postsurgical pain. Regional anaesthetic techniques are shown to improve outcomes such as postoperative analgesia, nausea, vomiting, delirium and promote early recovery. Currently majority of the breast cancer surgery is performed under general anaesthesia with a multimodal analgesic regimen with or without regional blocks. In fact, it is proved that breast cancer surgery can be done solely under regional anesthesia using multilevel thoracic paravertebral block (TPVB) with deep sedation, but rescue analgesia are often required intraoperatively, especially when surgeons handles the pectoralis muscle. Current evidence suggest that pectoral nerves, which are often described as a pure motor nerves that control movements only, also able to send noxious stimulation such as pain from the pectoral muscles and its deep fascia (via afferent nociceptive fibers) to the brain. Principal investigator proposes that adding a subpectoral plexus block (SPPB) will stop a wider spectrum of afferent nociceptive fibers from sending any pain signals than having thoracic paravertebral block alone. However, there is no report on the amount of local anaesthetic (LA) required to achieve surgical anaesthesia for breast surgery. The aim of this study is to evaluate the effectiveness of two different doses (10ml vs 20ml of 0.25% levobupivacaine) of local anaesthetic (LA) for subpectoral plexus in addition to 3 levels of TPVB injections at T2, T4, and T6 under ultrasound guidance for surgical anaesthesia for major breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for mastectomy, modified radical mastectomy or breast conservative surgery with lymph node biopsy and with or without axillary dissection

Exclusion Criteria:

* local skin site infection
* coagulopathy
* history of allergy to local anesthetics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients requiring intraoperative ketamine | during surgery
  The total number of patients (in percentage) requiring intraoperative ketamine bolus during the surgery

SECONDARY OUTCOMES:
Total amount of rescue ketamine used | during surgery
  The total amount of rescue ketamine (mg) required during surgery
Specific surgical region requiring rescue ketamine | during surgery
  The exact surgical region(s), such as infraclavicular, parasternal, axillary, subcostal) that rescue ketamine has to be given during surgery
Pain score on admission at Post Anaesthetic Care Unit (PACU) | Assessed once on admission at Post Anaesthetic Care Unit immediately after surgery
  Pain score (Numeric rating scale 0-100; 0=no pain, 100=severe pain) on admission at PACU
Pain score at Discharge of Post Anaesthetic Care Unit (PACU) | immediately before discharge from PACU
  Pain Score (Numeric rating scale 0-100; 0=no pain, 100=severe pain) at discharge from PACU

CONTACTS AND LOCATIONS:
Overall Officials: Manoj K Karmakar, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- North District Hospital, Sheung Shui, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No